CLINICAL TRIAL: NCT02503930
Title: The Effect of Transcranial Direct Cortical Stimulation (tDCS) on a Motor-cognitive Dual-task Performance of Parkinson's Patients
Brief Title: The Effect of tDCS on a Motor-cognitive Dual-task Performance of Parkinson's Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, michal roll, Director of Research and Development, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-15-NG-261-CTIL
Record Dates: First submitted 2015-07-09; First posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS (Experimental): The active tDCS condition will consist of 20 min of continuous stimulation. This amount of stimulation is safe for healthy young and older adults and has been shown to induce acute beneficial changes in cortical excitability and cognitive functions.
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): The Sham tDCS - an inactive stimulation.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — In this group subjects will receive 20 min of treatment.
  Other Names: Transcranial Direct Current Stimulation
  Arms: Active tDCS
Device: Sham tDCS — In this group subjects will receive 20 min of sham stimulation.
  Arms: Sham tDCS

SUMMARY:
The concurrent performance of two tasks, i.e., dual tasking (DT), is a common and ubiquitous every day phenomena. For example, people frequently walk while talking on a cellphone or drive while talking to a passenger. Often, the performance of one or more of these simultaneously performed tasks may deteriorate when another task is carried out at the same time, even in healthy young adults. This reduction in performance is referred to as the DT deficit or DT cost and is typically much higher in patients with Parkinson's disease (PD) than in young adults or age-matched controls. In PD, this DT cost impairs the gait pattern, as manifested, for example, in increased gait variability, exacerbating instability and fall risk.

In the proposed study, would be evaluated the effects of tDCS on dual tasking performance following tDCS.

The researchers expect that stimulation of the Pre Frontal Cortex (PFC) (using tDCS) will increase DT performance and prefrontal activation.

DETAILED DESCRIPTION:
tDCS intervention: Noninvasive tDCS will be delivered by study personnel uninvolved with any other study procedures. In the study will be used a battery-driven electrical stimulator. Stimulation and sham condition will be performed based on previous studies. Briefly, the anode will be placed over the PFC and the cathode over the right supraorbital region. The real tDCS condition will consist of 20 min of continuous stimulation at target intensity of 1.5 mA. This amount of stimulation is safe for healthy young and older adults and has been shown to induce acute beneficial changes in cortical excitability and cognitive functions. For the sham condition, an inactive stimulation protocol would be followed, as compared with an 'off-target' active protocol, in order to minimize participant risk. After each session, subjects will complete a side effects questionnaire. The efficacy of tDCS blinding will also be assessed after the final session, by asking each subject to judge whether they received real or sham tDCS, as well as their certainty of this judgment. Pre- and post-tDCS assessments will include:

fMRI: All of the MR images will be acquired on a 3.0 T scanner using an 8-channel head coil. T1-weighted brain volume (BRAVO) acquisitions will evaluate gray matter (GM) volume and thickness, markers of brain atrophy. This sequence will measure the ratio of GM within the PFC to overall GM, which will then be used to quantify the level of activation within the PFC. T2* echo planner imaging acquisition will be used for all the DT paradigms including intrinsic functional connectivity. Intrinsic connectivity will be examined while subjects are not engaged in any particular task and are requested to lie still with their eyes open (i.e., resting state). To examine task related changes versus more generalized patterns of DT activations, the type of the cognitive task or the nature of the motor task will be different in each task. The researchers will specifically examine the contribution of a secondary task involving working memory (arithmetic processing vs. attention), conflict monitoring, and motor planning on DT related activations.

fNIRS : fNIRS will be used to investigate the role of the frontal lobe in DT walking and how it is affected by tDCS [Mirelman et al. 2014]. The fNIRS system (Oxymon MKIII; Artinis Medical Systems) consists of flexible circuit board that carries the near-infrared light sources and detectors. The fNIRS sources and detectors pairs will be placed over the left (Fp1) and right (Fp2) frontal cortex regions of the forehead, as previously reported.

Gait assessment: Gait parameters will include both spatial and temporal parameters obtained using body fixed wearable sensors (accelerometers and gyroscopes) [Weiss et al. 2015;Ben et al. 2015]. Parameters will include (but are not limited to) gait speed, stride length and stride time as well as rhythmicity measures such as stride to stride variability and gait regularity.

The UPDRS, fall history and fear of falling will also be assessed (e.g., Falls Efficacy Scale International, FES-I) to further characterize the cohort and explore possible confounds.

Cognitive assessment: A detailed computerized cognitive battery that has been used extensively at TASMC in PD and other cohorts [Dwolatzky et al. 2003;Hausdorff et al. 2006;Springer et al. 2006;Yogev et al. 2005;Aarsland et al. 2003] will quantify several cognitive domains including working memory, executive function, verbal function, problem solving, a global cognitive score, and attention.

Sample size: Based on the effects of tDCS on DT walking outcomes in other cohorts [Leite et al. 2014;Zhou et al. 2014], the research group consider a conservative change of 15% in HbO2 levels after tDCS, as compared to sham, 18 subjects per group will provide >80% power. In order to allow for potential inter-subject variability and to address secondary questions (e.g., effect of disease severity), would be to assess 30 participants in each group.

Data collection:

A research assistant will assist participants filling in the electronic questionnaires and will conduct the non electronic ones (these would be later transcribed to excel sheets by research assistants).

A post-doc fellow and a PhD student will run the MRI scans and the tDCS sessions together with one-two research assistants. The participants will receive a reminder (by phone and or email) one day prior to each session. Participation will be monitored by the research assistants.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic PD (defined by the UK Brain Bank criteria)
2. Hoehn and Yahr score between 1.5-3
3. Taking anti-parkinsonian medications.

Exclusion Criteria:

1. Mini Mental State Exam (MMSE) score =< 24
2. Brain surgery in the past including implanted DBS
3. Major depression (DSM-IV Criteria)
4. Cerebral Infarction with Residual Deficits Diagnosis
5. Neurological diseases (except from PD)
6. Orthopaedic or cardiovascular diseases that may affect walking and cognitive abilities.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Changes in frequency and severity of the freezing of gait phenomenon | One week post intervention
  The new version of the Freezing of Gait questionnaire will be used to quantify the frequency and severity of this symptom. The score will be compared to baseline.

SECONDARY OUTCOMES:
fMRI scans - changes in gray matter (GM) volume | One week post intervention
  All of the MR images will evaluate gray matter (GM) volume, markers of brain atrophy.
fNIRS related frontal lobe activation - changes in tissue oxygenation | One week post intervention
  fNIRS will be used to investigate the role of the frontal lobe in DT walking and how it is affected by tDCS.The fNIR system provides with real-time monitoring of tissue oxygenation in the brain as subjects take different tests.
Changes in cognitive performance | One week post intervention
  The NeuroTrax software uses tests of cognitive performance that measure similar cognitive functions to traditional paper-based tests.
Immediate change in gait speed | One week post intervention
  Gait speed will be assessed under usual and dual task conditions and while negotiating physical obstacles, using a sensorized 7 meter carpet (PKMAS) and wearable body fixed sensors. These measures will be compared to baseline performance.
Immediate change in gait variability | One week post intervention
  Gait variability will be assessed under usual and dual task conditions and while negotiating physical obstacles, using a sensorized 7 meter carpet (PKMAS) and wearable body fixed sensors. These measures will be compared to baseline performance.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Giladi, M.D, Principal Investigator — Tel Aviv Sourasky medical Center, Tel Aviv, Israel. Phone: 972-3-6974790

REFERENCES:
- [Background] Zhou J, Hao Y, Wang Y, Jor'dan A, Pascual-Leone A, Zhang J, Fang J, Manor B. Transcranial direct current stimulation reduces the cost of performing a cognitive task on gait and postural control. Eur J Neurosci. 2014 Apr;39(8):1343-8. doi: 10.1111/ejn.12492. Epub 2014 Jan 20. PMID 24443958
- [Result] Leite J, Goncalves OF, Carvalho S. Facilitative effects of bi-hemispheric tDCS in cognitive deficits of Parkinson disease patients. Med Hypotheses. 2014 Feb;82(2):138-40. doi: 10.1016/j.mehy.2013.11.021. Epub 2013 Dec 1. PMID 24332532
- [Result] Springer S, Giladi N, Peretz C, Yogev G, Simon ES, Hausdorff JM. Dual-tasking effects on gait variability: the role of aging, falls, and executive function. Mov Disord. 2006 Jul;21(7):950-7. doi: 10.1002/mds.20848. PMID 16541455
- [Result] Weiss A, Herman T, Giladi N, Hausdorff JM. New evidence for gait abnormalities among Parkinson's disease patients who suffer from freezing of gait: insights using a body-fixed sensor worn for 3 days. J Neural Transm (Vienna). 2015 Mar;122(3):403-10. doi: 10.1007/s00702-014-1279-y. Epub 2014 Jul 29. PMID 25069586